CLINICAL TRIAL: NCT02235974
Title: Critical Periods After Stroke Study (CPASS); Sensitive Periods and Consumer Preferences: Optimizing Upper Extremity Stroke Rehabilitation
Brief Title: Critical Periods After Stroke Study (CPASS)
Acronym: CPASS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: MedStar National Rehabilitation Network (Other)
Collaborators: Georgetown University (Other); University of Wisconsin, Madison (Other); The Catholic University of America (Other); Medstar Health Research Institute (Other)
Responsible Party: Principal Investigator, Alexander W. Dromerick, MD, Vice President for Research, MedStar National Rehabilitation Network
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MNRH-2014-065
Record Dates: First submitted 2014-07-14; First posted 2014-09-10 (Estimated); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Stroke; Brain Infarction; Brain Ischemia; Cerebral Infarction; Cerebrovascular Disorders
Keywords: stroke; critical periods; sensitive periods; hemiparesis; upper extremity; physical rehabilitation; arm therapy; occupational therapy; physical therapy; task oriented training; patient focused; arm function; hand function; neurorehabilitation; motor learning; motor control; motor function; motor recovery; skill acquisition; skill training
MeSH Terms: conditions — Stroke; Brain Infarction; Brain Ischemia; Cerebral Infarction; Cerebrovascular Disorders; Paresis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Acute/Early (Experimental): Intervention: A 20-hour dose of early intensive upper extremity motor training therapy will be initiated within 30 days post-stroke.
  Interventions: Behavioral: Early Intensive upper extremity motor training
- Sub-acute/Outpatient (Experimental): Intervention: A 20-hour dose of sub-acute intensive upper extremity motor training therapy will be initiated within 2 to 3 months post-stroke.
  Interventions: Behavioral: Sub-acute intensive upper extremity motor training
- Chronic (Experimental): Intervention: A 20-hour dose of chronic intensive upper extremity motor training therapy will be initiated 6 to 9 months post-stroke
  Interventions: Behavioral: Chronic intensive upper extremity motor training
- Control (Placebo Comparator): Intervention: Usual and customary care. No additional therapy will be initiated during the 1-year study.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Early Intensive upper extremity motor training — Using a shaping therapy protocol, participants will receive a dose of 20 hours of intensive upper extremity therapy (in addition to their current therapy) beginning within 30 days of stroke onset.
  Arms: Acute/Early
Behavioral: Sub-acute intensive upper extremity motor training — Using a shaping therapy protocol, participants will receive a dose of 20 hours of intensive upper extremity therapy (in addition to their current therapy) beginning within 2 to 3 months post stroke.
  Arms: Sub-acute/Outpatient
Behavioral: Chronic intensive upper extremity motor training — Using a shaping therapy protocol, participants will receive a dose of 20 hours of intensive upper extremity therapy (in addition to their current therapy) beginning within 6 to 9 months post stroke.
  Arms: Chronic
Behavioral: Control — Usual and Customary Care only. No additional therapy will be given during the 1-year study.
  Arms: Control

SUMMARY:
To perform an exploratory single center randomized study that will form the basis for a larger scale, more definitive randomized clinical trial to determine the optimal time after stroke for intensive motor training. The investigators will perform a prospective exploratory study of upper extremity (UE) motor training delivered at higher than usual intensity at three different time points after stroke:

* early (initiated within 30 days)
* subacute/outpatient (initiated within 2-3 months)
* chronic (initiated within 6-9 months)

The control group will not receive the therapy intervention during the 1-year study.

Outcome measures will be assessed at baseline, pre-treatment, post-treatment, 6 months and one year after stroke onset.

Compared to individuals randomized during the outpatient (2-3 months after stroke onset) or chronic (6-9 months after stroke onset) time points, participants randomized to early intensive motor training will show greater upper extremity motor improvement measured at one year post stroke.

DETAILED DESCRIPTION:
Please see the following reference:

Dromerick, A.W., Edwardson, M., Edwards, D.F., Giannetti, M.L., Barth, J., Brady, K.P., Chan, E., Tan, M.T., Tamboli, I., Chia, R., Orquiza, M., Padilla, R.M., Cheema, A.K., Mapstone, M., Fiandaca, M.S., Federoff, H.J., & Newport, E.L. (2015). Critical Periods after Stroke Study: Translating animal stroke recovery experiments into a clinical trial. Frontiers in Human Neuroscience, 9, 002231. PMCID: PMC4413691.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic or hemorrhagic stroke (with confirmatory neuroimaging) within 28 days of admission to inpatient rehabilitation (allows those randomized to the early arm to begin study-related treatment within 30 days)
* Age >21 years
* Able to participate in first study-related treatment session within 30 days of stroke onset
* Able to participate in all study-related activities, including one year follow up and blood draws
* Persistent hemiparesis leading to impaired upper extremity function. Hemiparesis as indicated by NIHSS Motor Arm score ≥ 1
* Recovering moderate motor impairment at the shoulder and elbow or hand such as:

  * Proximal UE voluntary activity indicated by a score of ≥ 3 on the upper arm item of the Motor Assessment Scale - wrist and finger movement is not required

or

* Manual Muscle Test (MMT) score of ≥ 2 on shoulder flexion or abduction and MMT score of ≥ 2 for any of the following: elbow flexion, elbow extension, wrist flexion, wrist extension, finger flexion or finger extension.

or

* Active range of motion (AROM) to at least 50% of range in gravity eliminated position for shoulder flexion or abduction, and for any of the following motions: elbow flexion, elbow extension, wrist flexion, wrist extension, finger flexion or finger extension.

  * Score of ≤ 8 on the Short Blessed Memory Orientation and Concentration Scale
  * Follows 2 step commands
  * No upper extremity injury or conditions that limited use prior to the stroke
  * Pre-stroke independence: Modified Rankin Score 0 or 1

Exclusion Criteria:

* Inability to give informed consent
* Prior stroke with persistent motor impairment or other disabling neurologic condition such as multiple sclerosis, parkinsonism, amyotrophic lateral sclerosis (ALS), dementia requiring medication
* Rapidly improving motor function
* Clinically significant fluctuations in mental status in the 72 hours prior to randomization
* Hemispatial neglect as determined by >3 errors on the Mesulam Symbol Cancellation Test
* Not independent prior to stroke (determined by scores of <95 on Barthel Index or >1 on Modified Rankin Scale
* Dense sensory loss indicated by a score of 2 on NIHSS sensory item
* Ataxia out of proportion to weakness in the affected arm as described by a score of ≥ 1 on the NIHSS limb ataxia item
* Active or prior psychosis within 2 years
* Active or prior (within 2 years) substance abuse
* Not expected to survive 1 year due to other illnesses (cardiac disease, malignancy, etc)
* Received upper extremity botulinum toxin within 6 months (other medications do not exclude)

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2014-08-26 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-01-31 (Estimated)

PRIMARY OUTCOMES:
Action Research Arm Test (ARAT) | Baseline (within 30 days post stroke), pre-treatment, post-treatment (ideally within 72 hours after treatment has ended), 6 months and 1 year post stroke
  The ARAT assesses functional limitations and evaluates changes in limb function for the upper extremity.

SECONDARY OUTCOMES:
Motor Activity Log - 28 Quality of Movement (MAL-28 QOM) | Pre-treatment, post-treatment (ideally within 72 hours after treatment has ended), 6 months and 1 year post stroke
  A structured interview to measure upper extremity use and function as well as assess the quality of movement of the hemiparetic arm.
Nine Hole Peg Test (9-HPT) | Baseline (within 30 days post stroke), pre-treatment, post-treatment (ideally within 72 hours after treatment has ended), 6 months and 1 year post stroke
  A standardized quantitative test of upper extremity function and fine manual dexterity.
Functional Independence Measure (FIM) | Baseline (within 30 days post stroke), pre-treatment, post-treatment (ideally within 72 hours after treatment has ended), 6 months and 1 year post stroke
  A basic indicator of severity of disability. Tracks changes in the functional ability of the patient during an episode of hospital rehabilitation care.
Barthel Index (BI) | Baseline (within 30 days post stroke), pre-treatment, post-treatment (ideally within 72 hours after treatment has ended), 6 months and 1 year post stroke
  Measures performance in activities of daily living and functional disability.
Motricity Index - Arm only (MI) | Baseline (within 30 days post stroke), pre-treatment, post-treatment (ideally within 72 hours after treatment has ended), 6 months and 1 year post stroke
  To assess motor impairment and strength in the upper extremity.
Perception of change (POC) | Baseline (within 30 days post stroke), pre-treatment, post-treatment (ideally within 72 hours after treatment has ended) and 1 year post stroke
  A stroke-specific self-report to assess how stroke has impacted a person's life and their overall perception of recovery.
Stroke Impact Scale - Hand-Arm subscale (SIS) | Baseline (within 30 days post stroke), pre-treatment, post-treatment (ideally within 72 hours after treatment has ended) and 1 year post stroke
  A self-report health status measure to assess perceived recovery with regard to the more affected hand and arm following a stroke.
Modified Rankin Scale (MRS) | Baseline (pre-stroke assessment), pre-treatment, post-treatment (ideally within 72 hours after treatment has ended) and 1 year post stroke
  A measure of the degree of disability or dependence in daily activities following a stroke.
Activity Card Sort (ACS) | Pre-treatment (ideally within 72 hours of baseline), post-treatment (ideally within 72 hours after treatment has ended), 6 months and 1 year post stroke
  An interview-based assessment used to measure an individual's participation in instrumental, leisure and social activities.
Reintegration to Normal Living Index (RNLI) | Post-treatment (within 72 hours after treatment has ended), 6 months and 1 year post stroke
  To assess quantitatively the degree that individuals who have experienced a traumatic injury or illness come to manage and reintegrate normal social activities with regard to recreation, movement at home and within the community, family and relationships.
Geriatric Depression Scale (GDS-15) | Baseline (within 30 days post stroke), pre-treatment, and 1 year post stroke
  A self-report assessment used to identify depressive symptoms in the elderly.
NIH Stroke Scale (NIHSS) | Baseline (within 30 days post stroke), pre-treatment, 6 months and 1 year post stroke
  A systematic assessment used to evaluate and measure stroke-related. neurological impairments and stroke severity.
Short Blessed Orientation and Memory Concentration Test (SBT) | Baseline (within 30 days post stroke)
  An assessment of cognitive ability and impairment.
Mesulam Symbol Cancellation Test (SCT) | Baseline (within 30 days post stroke)
  An assessment used to evaluate visuospatial function and attention.
Faces Pain Scale | Baseline (within 30 days post stroke), pre-treatment, post-treatment (ideally within 72 hours after treatment has ended), 6 months and 1 year post stroke
  A self-report measure of pain intensity.
Fugl Meyer Assessment (Upper Extremity) | Baseline (within 30 days post stroke) and 1 year post stroke
  A performanced-based impairment index to assess motor function, sensation and joint function.
Manual Muscle Test (Upper Extremity) | Baseline (within 30 days post stroke)
  Muscle strength assessment

OTHER OUTCOMES:
Motor Assessment Scale - Upper Arm Function (MAS) | Baseline (within 30 days of stroke onset)
  Performance-based scale to assess everyday motor function.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander W Dromerick, MD, Principal Investigator — MedStar National Rehabilitation Network
Locations (1):
- MedStar National Rehabilitation Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan at this time to make individual participant data available.

REFERENCES:
- [Background] Dromerick AW, Edwardson MA, Edwards DF, Giannetti ML, Barth J, Brady KP, Chan E, Tan MT, Tamboli I, Chia R, Orquiza M, Padilla RM, Cheema AK, Mapstone ME, Fiandaca MS, Federoff HJ, Newport EL. Critical periods after stroke study: translating animal stroke recovery experiments into a clinical trial. Front Hum Neurosci. 2015 Apr 29;9:231. doi: 10.3389/fnhum.2015.00231. eCollection 2015. PMID 25972803
- [Derived] Geed S, Feit P, Edwards DF, Dromerick AW. Why Are Stroke Rehabilitation Trial Recruitment Rates in Single Digits? Front Neurol. 2021 Jun 8;12:674237. doi: 10.3389/fneur.2021.674237. eCollection 2021. PMID 34168611